CLINICAL TRIAL: NCT05718843
Title: Pharmacokinetics, Safety and Tolerability of BI 425809 (Iclepertin) Following Oral Administration in Male and Female Participants With Different Degrees of Renal Impairment (Severe, Moderate and Mild) Compared With Matched Male and Female Participants With Normal Renal Function (an Open-label, Non-randomised, Single-dose, Parallel, Individual-matched Design Trial)
Brief Title: A Study to Test How Iclepertin is Taken up in the Blood of People With and Without Kidney Problems
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1346-0047; 2022-002739-74 (EudraCT Number)
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — BI 425809

STUDY DESIGN:
Intervention Model Description: Non-randomised, single dose, open-label, individual-matched design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1: Participants with severe renal impairment (Experimental)
  Interventions: Drug: BI 425809
- Group 2: Participants with normal renal function individually matched to participants of Group 1 (Experimental)
  Interventions: Drug: BI 425809
- Group 3: Participants with moderate renal impairment (Experimental)
  Interventions: Drug: BI 425809
- Group 4: Participants with normal renal function matching Group 3 (Experimental)
  Interventions: Drug: BI 425809
- Group 5: Participants with mild renal impairment (Experimental)
  Interventions: Drug: BI 425809
- Group 6: Participants with normal renal function matching Group 5 (Experimental)
  Interventions: Drug: BI 425809

INTERVENTIONS:
Drug: BI 425809 — BI 425809
  Other Names: Iclepertin

SUMMARY:
This study is open to people with and without kidney problems. People can join the study if they are 18 years or older and have a body mass index (BMI) between 18.5 and 35 kg/m2.

Iclepertin is a medicine that is being developed to treat diseases of the brain. The purpose of this study is to find out whether having kidney problems influences how iclepertin is taken up in the body. All participants take iclepertin once as a tablet.

Participants are in the study for 2 to 3 weeks. During this time, they visit the study site 6 times. For one of the visits, participants stay 4 nights at the study site. The site staff measures the amount of iclepertin in the blood. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria applicable to all participants

* Male or female participants
* Age of at least 18 years (inclusive)
* BMI of 18.5 to 35 kilogram per square metre (kg/m2) (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) - Good Clinical Practice (GCP) and local legislation prior to admission to the trial
* Male participants are not required to use contraception
* Woman of childbearing potential (WOCP) are allowed to participate provided they use a highly effective contraception from at least 30 days before the administration of trial medication until 30 days after trial completion. The following methods of contraception are considered adequate for female participants of childbearing potential:

  * Use of combined (oestrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal), plus condom
  * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus condom
  * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
  * Sexually abstinent
  * A vasectomised sexual partner who received medical assessment of the surgical success (documented absence of sperm) and provided that partner is the sole sexual partner of the trial participant.

Female participants are not considered to be of childbearing potential if they are either surgically sterilised (including hysterectomy) or postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of Follicle-stimulating hormone (FSH) above 40 Units per Litre (U/L) and oestradiol below 30 nanogram per Litre (ng/L) is confirmatory)

Inclusion criteria applying only to participants with impaired renal function

* Renal impairment based on assessment of estimated Glomerular Filtration Rate (eGFR) at screening (severe renal impairment: 15-29 millilitre per minute per 1.73 square metre (mL/min/1.73 m2), moderate renal impairment: 30-59 mL/min/1.73 m2, mild renal impairment: 60-89 mL/min/1.73 m2)
* Chronic renal impairment > 12 months (documented renal impairment indicated by reduced eGFR for more than 12 months until screening)
* Absence of clinically significant abnormalities, as based on a complete medical history including a full physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests at both screening and check-in, with the exception of findings that in the opinion of the investigator are consistent with the participant's renal impairment
* Medication and/or treatment regimens must have been stable (i.e., no dose adjustments) for at least 4 weeks prior to the screening period and should be kept stable until study completion. Fluctuating treatment regimens may be considered for inclusion on a case-by-case basis if the underlying disease is under control in the opinion of the investigator and must be agreed to by both the investigator and the sponsor's medical monitor

Inclusion criteria applying only to participants with normal renal function

* Individually matched to participants with renal impairment according to sex, age, and weight, and race
* eGFR ≥ 90 mL/min/1.73 m2
* Absence of clinically significant abnormalities identified by a detailed medical history, full physical examination, vital signs and 12-lead ECG at both screening and check-in visits
* Absence of clinically significant abnormalities identified by a laboratory test at screening visit

Exclusion criteria applying to all participants

* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics (PK) of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the Central Nervous System (CNS) (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders (including but not limited to major depressive disorder)
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Relevant chronic or acute infections
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days (or 5 of its half-lives, whichever is longer) of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause ECG interval from the start of the QRS complex to the end of the T wave (QT interval) / QT interval corrected for heart rate, e.g. using the method of Fridericia (QTcF) or Bazett (QTcB) (QTc interval) prolongation ) Further exclusion criteria apply.

Exclusion criteria applying only to participants with renal impairment

* A marked prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 480 milliseconds (ms) in males or repeatedly greater than 500 ms in females) or any other relevant ECG finding at screening
* Acute renal failure or active nephritis
* Nephrotic syndrome
* Impaired hepatic function, including relevant increases in liver enzymes indicating liver disease
* Relevant diseases for which it can be assumed that the absorption of the study drugs will not be normal (i.e., relevant malabsorption, chronic diarrhoea)
* Participant under dialysis or planned to start dialysis during participation in the study
* History of myocardial infarction, cerebrovascular accident or severe arrhythmia within the 6 months prior to the screening visit.
* History of vascular surgery or intervention (e.g., coronary artery bypass, percutaneous transluminal angioplasty etc.) less than 6 months prior to dosing Further exclusion criteria apply.

Exclusion criteria applying only to participants with normal renal function

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* A marked prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant ECG finding at screening
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg) (for participants older than 60 years: 90 to 150 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 (beats per minute) bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of BI 425809 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Up to 7 days.
Maximum measured concentration of BI 425809 in plasma (Cmax) | Up to 7 days.

SECONDARY OUTCOMES:
Area under the concentration-time curve of BI 425809 in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf) | Up to 7 days.

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com